CLINICAL TRIAL: NCT05473494
Title: THE EFFECT OF ONLINE TRAININGS ON DIABETIC FOOT CARE ON FOOT CARE BEHAVIOR AND SELF-EFFECTIVENESS ATTITUDES OF INDIVIDUALS WITH TYPE II DIABETES
Brief Title: THE EFFECT OF ONLINE TRAINING ON FOOT CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Ayşegül Kandemir, Principal Investigator, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021/33-03
Record Dates: First submitted 2022-06-22; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Type2diabetes; Diabetic Foot
Keywords: Type2diabetes; DiabeticFootCare; OnlineEducational; DistanceEducation; Self-Effectıveness
MeSH Terms: conditions — Diabetic Foot | interventions — Sensitivity Training Groups; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Experimental)
  Interventions: Other: training group
- control group (Active Comparator)
  Interventions: Other: control group

INTERVENTIONS:
Other: training group — Trainings on diabetic foot care consisting of min 20 max 40 minutes will be given in 5 sessions for nine weeks. Training will be given face to face online.
  Arms: training group
Other: control group — Group not to be trained.
  Arms: control group

SUMMARY:
The aim of this study is to determine the effect of online trainings on diabetic foot care on foot care behavior and self-efficacy attitudes of individuals with type II diabetes.

Purpose in accordance with the patient's Diagnostic Information Form, diabetic foot care self-efficacy Scale(DABOO), foot care Behavior Scale(ABDO) and diabetic foot risk screening forms are available in the data collection tools; education and Research Hospital Internal Medicine outpatient clinic with Deeply Izmit Seka state hospital, inpatient or outpatient treatment for persons with Type II diabetes who agree to volunteer to participate in research 90 shall apply. After that, the groups will be divided into two groups by randomization, and one of the groups will be given training sessions consisting of min 20 max 40 minutes for diabetic foot care in 5 sessions for nine weeks. After the training, the scales will be applied to the groups again. The data obtained before and after the training will be compared statistically in a computer environment

ELIGIBILITY:
Inclusion Criteria:

* Patients who were applied the Dietetic Foot Risk Screening form during the physician's examination and who were in the low and medium risk groups after the physician's examination.
* To be able to read and write.
* Being between the ages of 18-65.
* Being on oral antidiabetic (OAD) and/or insulin therapy.
* No restriction of access to the Internet.
* To be able to use the Zoom program or WhatsApp video conversation with or without support.
* Having computer and/or telephone skills.
* Volunteering to participate in the study (Informed consent form will be signed by the participants during the application)
* Not having sensory loss such as speech and hearing that prevents communication and no psychiatric problems.

Exclusion Criteria:

outside the inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-25 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Diabetic Foot Care Self-Efficacy Scale | nine weeks
  Self-efficacy is measured by scoring between 0 and 10. The 9 expressions that make up the scale are evaluated on the 11-digit visual scale, which is specified as -Not sure=0 and very sure=10. The lowest score of the scale is 0 and the highest score is 100. As the score obtained from the scale increases, the diabetic foot self-efficacy level increases in parallel.

SECONDARY OUTCOMES:
Foot Care Behavıor Scale | nine weeks
  Consisting of 15 items in a 5-point Likert type, the scale is scored according to agree-disagree (1= Never, 2= Occasionally, 3= Sometimes, 4= Often, and 5= Always) and consists of 15 items. The lowest score that can be obtained from the scale, which evaluates foot care behavior as a single dimension, is 15 and the highest score is 75. An increase in the scale score indicates that the individual's foot self-care behaviors become positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Ev, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No